CLINICAL TRIAL: NCT02088905
Title: Efficacy of Parent-Child Interaction Therapy With ASD
Brief Title: Efficacy of Parent-Child Interaction Therapy With Autism Spectrum Disorder
Acronym: PCIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Benjamin L Handen, PhD, BCBA-D, Assoicate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0031588; PRO023120445 (Other: University of Pittsburgh IRB)
Record Dates: First submitted 2014-03-07; First posted 2014-03-17 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Noncompliance
Keywords: PCIT, autism, parent training, noncompliance
MeSH Terms: conditions — Patient Compliance; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent Child Interaction Therapy (Experimental): Families will either receive Parent Child Interaction Therapy or be placed on a wait-list control group
  Interventions: Behavioral: Parent Child Interaction Therapy
- Wait list control (No Intervention): Families will wait 18 weeks for treatment, serving as controls.

INTERVENTIONS:
Behavioral: Parent Child Interaction Therapy — Parent-Child Interaction Therapy (PCIT) is a research-supported parent coaching intervention that has been found to be highly effective among typically developing preschoolers presenting with a range of mental health concerns, especially defiance and noncompliance.6 PCIT holds considerable promise as a potentially effective treatment for children with ASD because it directly addresses the behaviors parents of children with ASD report to be most problematic for them - defiance, stubbornness, and temper tantrums. PCIT is theoretically consistent with other approaches that have shown promise in treating ASD (i.e., behaviorally-based); however, PCIT is unique in that it incorporates a socially-based initial phase which may have some unique benefits for children with ASD.
  Arms: Parent Child Interaction Therapy

SUMMARY:
The aim of the current proposal is to determine if the PCIT treatment manual can be successfully utilized for preschoolers with ASD and disruptive behavior (across a range of intellectual functioning levels) and to evaluate its ability to significantly decrease measures of problem behavior. It is hypothesized that the current manual will require few modifications for use with ASD and that, in comparison to a wait-list control group, families who undergo PCIT training will evidence significant gains on measures of parenting stress, child externalizing behaviors and compliance to parental requests. To address the pilot study aims, we will recruit a total of 25 families of children with ASD (ages 2.6-6.11 years) whose children are already receiving intensive, one-on-one behavioral treatment services (15-30 hours per week) but no structured parent training. Families will be randomized to either intensive services + PCIT or intensive services alone (wait list control). Assessments will be completed at baseline, mid-treatment (9 weeks post baseline), post-treatment (18 weeks after the baseline assessment) and long-term follow-up (12 weeks post-treatment). PCIT families will attend 16 weekly, one-hour coaching sessions. Both active treatment and wait-list control families will continue to receive intensive ABA services in the home or community. Control families will receive PCIT training after 18 weeks on the "wait-list." The aims of the pilot study are:

1. To assess the utility of the current PCIT treatment manual with preschoolers with ASD and disruptive behavior and their parents;

   Hypothesis 1: The current PCIT treatment manual will be able to be utilized with families of children with ASD with only minimal modifications.

   Hypothesis 2: Families of children with ASD will consistently attend PCIT sessions.
2. To determine if PCIT with this population will result in an increase in appropriate parent behaviors and a subsequent decrease in targeted child behaviors (e.g., direct assessment of noncompliance, behavior rating scales).

Hypothesis 3: Families receiving PCIT training will evidence statistically greater decreases on measures of disruptive behavior, quality of parent-child interactions and parental stress than families on the wait-list control group.

DETAILED DESCRIPTION:
Young children with ASD often present with a range of externalizing behavior problems, including aggression, tantrums and difficulty transitioning. Interventions based on the principles of applied behavior analysis (ABA) have been shown to offer an effective means of addressing many of these concerns. Parent-Child Interaction Therapy (PCIT) is a manualized, empirically supported parent coaching intervention that has been found to be highly effective for typically developing preschoolers presenting with a range of mental health concerns. It also holds considerable promise as a potentially effective treatment for children with ASD. The focus of PCIT treatment is to both improve parent-child interactions and to reduce child behavior problems. PCIT involves the coaching of parents in real-time, via a one-way mirror and a "bug-in-the ear" device that allows the therapist to provide feedback and directions to the parent while interacting with his/her child. The aim of the current proposal is to determine if the PCIT treatment manual can be successfully utilized for preschoolers with ASD and to evaluate its ability to significantly decrease measures of problem behavior. It is hypothesized that the current manual will require few modifications for use with ASD and that, in comparison to a wait-list control group, families who undergo PCIT training will evidence significant gains on measures of parenting stress, child externalizing behaviors and compliance to parental requests. To address the pilot study aims, we will recruit a total of 25 families of children with ASD (ages 2.6-6 years) whose children are already receiving intensive, one-on-one behavioral treatment services (15-30 hours per week). Families will be randomized to either intensive services + PCIT or intensive services alone (wait list control). Assessments will be completed at baseline, mid-treatment (9 weeks post baseline) and post-treatment (18 weeks after the baseline assessment). PCIT families will attend 20 weekly, one-hour coaching sessions. Both active treatment and wait-list control families will continue to receive intensive ABA services in the home or community. The results of this study will provide pilot data in a subsequent application for federal funding to conduct larger controlled trials, including examining the use of PCIT in school-age children with ASD and intellectual disability and to assess the individual and combined efficacy of PCIT and psychopharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

i. Outpatients between 2 years, 6 months and 6 years, 11 months of age; ii. Diagnosis of Autistic Disorder, Pervasive Developmental Disorder Not Otherwise Specified, or Asperger's Disorder based upon the Autism Diagnostic Observation Schedule and clinical evaluation by Diagnostic and Statistical Manual of Mental Disorders IV criteria; iii. Males and females; iv. Mental Age>30 months based upon the Stanford-Binet V or Mullens [to insure that the child possesses enough expressive language to offer opportunities for the parent to learn "verbal reflection" skills and that child is able to understand time out]; v. Eyberg Child Behavior Inventory score greater than or equal to 120; vi. Behavior Assessment System for Children Externalizing Problem Scale T-score >65; vii. Care provider who can reliably bring subject to clinic visits, can attend weekly PCIT sessions, can provide trustworthy ratings and interact with subject on a regular basis.

Exclusion Criteria:

i. Unstable use of psychotropic medications (no changes in dose for at least two months and no plans to change dose during the course of the study); ii. Unstable use of dietary supplements (e.g., casein-gluten free diet)(no changes in supplement dose for at least two months and no plans to change douse during the course of the study); iii. Prior involvement in PCIT or currently receiving parent training. iv. Extremely severe behavioral concerns that require immediate treatment

Ages: 30 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Handen, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Merck Child Outpatient Clinic, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began June 2014, with clinicians at the Merck Center for Autism and Developmental Disorders or from the Child Development Unit bringing up the study to patients.
  140 subjects were excluded during phone screen. 77 did not meet inclusion criteria, 39 declined consent due to high burden of time/procedures, 24 refused for other reasons.
Pre-assignment Details: Two subjects of the originally enrolled 25 were discovered to have not met inclusion criteria. Upon the discovery, they were removed from the study and not randomized to any study condition.
Period: Overall Study
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Started | 13 | 10
Week 9 (Last Observation Carried Forward for 10 treatment and 9 wait list who completed Week 9 Assessment) | 10 | 9
Completed (Last Observation Carried Forward for 10 treatment and 9 wait list who completed Week 9 Assessment) | 8 | 9
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Parent Child Interaction Therapy: Families will either receive Parent Child Interaction Therapy or be placed on a wait-list control group
  Parent Child Interaction Therapy: Parent-Child Interaction Therapy (PCIT) is a research-supported parent coaching intervention that has been found to be highly effective among typically developing preschoolers presenting with a range of mental health concerns, especially defiance and noncompliance.6 PCIT holds considerable promise as a potentially effective treatment for children with Autism Spectrum Disorder because it directly addresses the behaviors parents of children with ASD report to be most problematic for them - defiance, stubbornness, and temper tantrums. PCIT is theoretically consistent with other approaches that have shown promise in treating ASD (i.e., behaviorally-based); however, PCIT is unique in that it incorporates a socially-based initial phase which may have some unique benefits for children with ASD.
- Total: Total of all reporting groups
Arm/Group | Parent Child Interaction Therapy | Wait List Control | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: months] — Child's age at the beginning of the study
  months | 63.62 (17.08) | 67.0 (16.31) | 65.087 (16.45631)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Caucasian | 11 | 10 | 21
  Hispanic | 0 | 0 | 0
  Native American | 0 | 0 | 0
  Mixed Race | 0 | 0 | 0
Peabody Picture Vocabulary Test [Mean (Standard Deviation); unit: units on a scale] — Peabody Picture Vocabulary Test Raw Score - IV PPVT-IV is a test for a child's receptive vocabulary, with higher scores indicating greater verbal ability and scholastic skills. Range for the raw score is 20-160. Population: Missing data for one participant
  units on a scale
    number analyzed (Participants) | 12 | 10 | 22
    (all) | 97.83 (13.27) | 105.20 (16.24) | 101.18 (14.81)
Intelligence Quotient (IQ) [Mean (Standard Deviation); unit: units on a scale] — A full scale intelligence quotient (IQ) score provided by the Stanford-Binet Intelligence Scales, K-SEALS, WPPSI-IV.
  IQ tests have range of 0-200. Higher IQ scores from any measure indicate greater cognitive capacity with 90-109 considered average.
  units on a scale | 93.38 (15.68) | 103.60 (21.29) | 97.83 (19.02)
Parental Stress Index [Mean (Standard Deviation); unit: units on a scale] — Parental Stress Index-4 Short Form (PSI):Total Stress Scale, total of subscales, range 36-180, higher indicating more parental stress. Defensive Responding, range 7 - 35. Lower scores indicate higher defensive responding from parents. Parental Distress, range 12- 60. Higher scores indicate more parental stress. Parent-Child Dysfunctional Interaction subscale, range 12 - 60. Higher scores indicate parents feel their child is not meeting their expectations when interacting. Difficult Child, range is 12 - 60. Higher scores indicate that parents view their child to be difficult to parent.
  units on a scale
    PSI Defensive Responding | 19.62 (5.55) | 19.30 (6.88) | 19.48 (6.01)
    Parent Distress Subscale Score | 32.31 (9.38) | 31.30 (10.25) | 31.87 (9.56)
    Parent-Child Dysfunctional Interaction Subscale Sc | 32.54 (7.58) | 28.80 (8.68) | 30.91 (8.11)
    Difficult Child Subscale Score | 43.15 (5.71) | 40.80 (6.83) | 42.13 (6.19)
    Total Stress | 108.00 (18.75) | 101.00 (22.32) | 104.96 (20.20)
Eyberg Child Behavior Inventory [Mean (Standard Deviation); unit: units on a scale] — Eyberg Child Behavior Inventory (ECBI):
  Intensity score range is 36 - 252, with higher scores indicating a higher frequency of problem behaviors.
  The ECBI contains the Problem Score calculated from 36 items rated on whether the particular behavior is considered by the to be a problem (yes) or not (no).
  Problem score range is from a minimum of 0 - 36, with higher scores indicating more behaviors that a parent considers to be a problem.
  units on a scale
    Intensity | 166.00 (29.8) | 157.30 (21.0) | 162.22 (26.1)
    Problem | 19.46 (8.56) | 20.00 (5.66) | 19.70 (7.29)
Dyadic Parent-Child Interaction Coding [Mean (Standard Deviation); unit: Frequency of Behavior] — The Dyadic Parent-Child Interaction Coding System (DPICS) codes frequency of behaviors that occur during five minutes of child lead play, then parent lead play, and then clean-up.
  Positive Skills was the total frequency of behavioral descriptions, reflections, and labeled praise throughout the three conditions.
  Negative skills score was a combination of the total frequency of questions and negative talk throughout all conditions, as well as total commands during child lead play. It was expected that parent would give commands during parent-lead play or clean-up. Population: Data missing for one participant
  Frequency of Behavior
    Positive Skills: number analyzed (Participants) | 12 | 10 | 22
    Positive Skills | 6.67 (4.23) | 8.30 (6.13) | 7.41 (5.11)
    Negative Skills: number analyzed (Participants) | 12 | 10 | 22
    Negative Skills | 73.92 (21.66) | 97.10 (27.60) | 84.45 (26.68)
Social Responsiveness Scale 2 [Mean (Standard Deviation); unit: units on a scale] — Social Responsiveness Scale 2nd edition (SRS-2). SRS-2 Total Score is sum of subscales, for all subscales, higher scores mean more impairment. Total score range is 0-195. Social Awareness measures social awareness impairment, range 0-24. Social Cognition measures social cognition impairment, range 0-36. Social Communication measures social communication impairment, range 0-66. Social Motivation measures social motivation impairment, range 0-33. Restricted and Repetitive Behaviors measures restricted and repetitive behaviors, range 0-36.
  units on a scale
    SRS Total Raw Score | 99.08 (24.65) | 88.30 (21.74) | 94.39 (23.55)
    SRS Awareness Raw Score | 13.62 (2.75) | 12.20 (3.77) | 13.00 (3.23)
    SRS Cognition Raw Score | 17.92 (5.96) | 15.10 (3.54) | 16.70 (5.16)
    SRS Communication Raw Score | 32.15 (10.47) | 30.40 (7.86) | 31.39 (9.27)
    SRS Motivation Raw Score | 16.38 (4.86) | 12.20 (3.68) | 14.57 (4.78)
    SRS Restricted and Repetitive Behaviors Raw Score | 19.00 (7.44) | 18.40 (7.07) | 18.74 (7.12)

OUTCOME MEASURES:

1. Primary Outcome: Eyberg Child Behavior Inventory
Description: Eyberg Child Behavior Inventory (ECBI). For families receiving PCIT training, the ECBI will be completed at screen, at each PCIT training visit and at the 12-week post-treatment visit. Wait-list control families will complete the ECBI at screen as well as at weeks 9 and 18. Reported week 9.
  The ECBI contains the Intensity Score calculated from 36 items rated on frequency of behavior from 1 (Never) to 7 (Always).
  Intensity score range is 36-252, with higher scores indicating a higher frequency of problem behaviors.
  The ECBI contains the Problem Score calculated from 36 items rated on whether the particular behavior is considered by the to be a problem (yes) or not (no).
  Problem score range is 0-36, with higher scores indicating a higher frequency of problem behaviors.
Time Frame: Week 9
Population: Subjects who dropped out prior to Week 9 (2 in treatment group, 1 in wait list control) were not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
units on a scale
  ECBI Intensity Score | 132.50 (42.62) | 154.33 (25.60)
  ECBI Problem Score | 18.9 (9.65) | 19.11 (6.45)

2. Primary Outcome: Eyberg Child Behavior Inventory
Description: Eyberg Child Behavior Inventory (ECBI). For families receiving PCIT training, the ECBI will be completed at screen, at each PCIT training visit and at the 12-week post-treatment visit. Wait-list control families will complete the ECBI at screen as well as at weeks 9 and 18. Reported week 18
  The ECBI contains the Intensity Score calculated from 36 items rated on frequency of behavior from 1 (Never) to 7 (Always).
  Intensity score range is 36-252, with higher scores indicating a higher frequency of problem behaviors.
  The ECBI contains the Problem Score calculated from 36 items rated on whether the particular behavior is considered by the to be a problem (yes) or not (no).
  Problem score range is 0-36, with higher scores indicating a higher frequency of problem behaviors.
Time Frame: Week 18
Population: Following the intent-to-treat principle, last observation carried forward for 2 subjects in treatment group who dropped out after Week 9. Subjects who dropped out prior to Week 9 (2 in treatment group, 1 in wait list control) were not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
units on a scale
  ECBI Intensity Score | 115.20 (41.54) | 148.67 (25.25)
  ECBI Problem Score | 14.10 (10.54) | 19.67 (5.00)
Statistical Analysis 1: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of ECBI Problem Score between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .080, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of ECBI Intensity Score between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .026, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Parent Child Interaction Therapy vs Wait List Control; Mixed Model Analysis of ECBI Intensity Scores, with variables of Timepoint, Treatment Assignment, and Timepoint*Treatment Assignment interaction. Random intercept used; Test type: Other — Type III Tests of Fixed Effects; p < .001, Mixed Models Analysis — Mixed Model Analysis - Significance of Timepoint within the model in determining the effectiveness of assigned treatment
Statistical Analysis 4: Comparison: Parent Child Interaction Therapy vs Wait List Control; [analysis description as in outcome 2, analysis 3]; Test type: Other — Type III Tests of Fixed Effects; p = .182, Mixed Models Analysis — Mixed Model Analysis - Significance of Treatment Assignment within the model in determining the effectiveness of assigned treatment
Statistical Analysis 5: Comparison: Parent Child Interaction Therapy vs Wait List Control; [analysis description as in outcome 2, analysis 3]; Test type: Other — Type III Tests of Fixed Effects; p = .015, Mixed Models Analysis — Mixed Model Analysis - Significance of Treatment Assignment and Timepoint Interaction Term within the model in determining the effectiveness of assigned treatment

3. Secondary Outcome: Parental Stress Index-4 Short Form
Description: Parental Stress Index-4 Short Form (PSI) is comprised of several subscales that are independently measured and also combined to create a total score. Scores are calculated from 36 questions that rated as Strongly Agree/Agree/Not Sure/Disagree/Strongly Disagree by the parents. Ratings are attached to a 5-point Likert scale.
  PSI Defensive Responding subscale range: 7-35. Lower scores indicate higher defensive responding from parents.
  For the PSI Parental Distress subscale, range 12-60. Higher scores indicate higher parental stress in the parenting.
  For the PSI Parent-Child Dysfunctional Interaction subscale, range 12-60. Higher scores indicate parents feel their child is not meeting their expectations when interacting.
  For the PSI Difficult Child subscale, range 12-60. Higher scores indicates parents view their child to be difficult to parent.
  For PSI Total Stress, range 43-215. Higher scores indicate higher stress.
Time Frame: Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
units on a scale
  PSI Defensive Responding | 17.70 (7.21) | 20.33 (4.77)
  Parent Distress Subscale Score | 29.10 (12.28) | 33.44 (9.53)
  Parent-Child Dysfunctional Interaction Subscale | 28.80 (7.98) | 27.44 (7.32)
  Difficult Child Subscale Score | 38.20 (12.59) | 43.56 (5.50)
  Total Stress | 96.10 (28.67) | 104.56 (18.21)
Statistical Analysis 1: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of PSI Parental Distress between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .203, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of PSI Parent-Child Dysfunctional Interaction between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of PSI Difficult Child between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = 0.308, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of PSI Total Score between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .413, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons

4. Secondary Outcome: Social Responsiveness Scale 2 Score
Description: Social Responsiveness Scale 2nd edition (SRS-2). SRS-2 Total Score is sum of subscales, higher scores mean more impairment. Range 0-195. Social Awareness measures social awareness impairment, higher scores mean more impairment. Range 0-24. Social Cognition measures social cognition impairment, higher scores mean more impairment. Range 0-36. Social Communication measures social communication impairment, higher scores mean more impairment. Range 0-66. Social Motivation measures social motivation impairment, higher scores means more impairment. Range 0 - 33. Restricted and Repetitive Behaviors measures restricted and repetitive behaviors, with higher scores indicating more impairment. Range 0 - 36.
Time Frame: Week 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
units on a scale
  Total Raw Score | 91.20 (34.31) | 92.22 (17.65)
  Awareness Raw Score | 13.20 (3.19) | 12.78 (2.11)
  Cognition Raw Score | 15.80 (7.30) | 16.00 (3.04)
  Communication Raw Score | 30.80 (13.31) | 32.78 (7.58)
  Motivation Raw Score | 14.40 (5.74) | 12.22 (3.38)
  Restricted and Repetitive Behaviors Raw Score | 17.00 (8.71) | 18.44 (7.21)

5. Secondary Outcome: Social Responsiveness Scale 2 Score
Description: as for outcome 4
Time Frame: Week 18
Population: Data missing from some participants. Following the intent-to-treat principle, last observation carried forward for 2 subjects in treatment group who dropped out after Week 9. Subjects who dropped out prior to Week 9 (2 in treatment group, 1 in wait list control) were not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
units on a scale
  Total Raw Score | 80.00 (28.25) | 88.22 (29.12)
  Awareness Raw Score | 12.40 (2.67) | 12.11 (4.65)
  Cognition Raw Score | 14.60 (5.97) | 15.89 (4.08)
  Communication Raw Score | 27.10 (10.26) | 30.67 (11.25)
  Motivation Raw Score | 11.10 (5.38) | 11.44 (4.59)
  Restricted and Repetitive Behaviors Raw Score | 14.80 (8.38) | 18.11 (8.54)
Statistical Analysis 1: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of SRS Total Score between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = 0.271, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of SRS Awareness Score between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .434, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of SRS Cognition Scores between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .298, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of SRS Communication Score between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .294, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of SRS Motivation between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .441, t-test, 1 sided — No adjustment for multiple comparisons
Statistical Analysis 6: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of SRS Restricted and Repetitive Behavior Score between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p = .204, t-test, 1 sided — No adjustment for multiple comparisons

6. Secondary Outcome: Dyadic Parent-Child Interaction Coding System Scores
Description: The Dyadic Parent-Child Interaction Coding System (DPICS) codes frequency of behaviors that occur during five minutes of child-lead play, then parent-lead play, and then clean-up.
  Positive Skills score is the total frequency of behavioral descriptions, reflections, and labeled praise throughout the three conditions.
  Negative skills score is a combination of the total frequency of questions, negative talk, and indirect commands throughout all conditions, as well as direct commands during child lead play. It was expected that parents would give commands during parent-lead play or clean-up.
Time Frame: Week 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: frequency of behaviors
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
frequency of behaviors
  Negative Skills | 35.2 (14.54) | 81.78 (19.886)
  Positive Skills | 26.9 (16.28) | 5.667 (5)

7. Secondary Outcome: Dyadic Parent-Child Interaction Coding System Scores
Description: The Dyadic Parent-Child Interaction Coding System (DPICS) codes frequency of behaviors that occur during five minutes of child lead play, then parent lead play, and then clean-up.
  Positive Skills score was the total frequency of behavioral descriptions, reflections, and labeled praise throughout the three conditions.
  Negative skills score was a combination of the total frequency of questions, negative talk, and indirect commands throughout all conditions, as well as direct commands during child lead play. It was expected that parents would give commands during parent-lead play or clean-up.
Time Frame: Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: counts of behaviors
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
counts of behaviors
  Negative Skills | 22.2 (14.71) | 76.44 (24.6)
  Positive Skills | 41.4 (23.98) | 8.11 (6.29)
Statistical Analysis 1: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of DPICS Negative Skills between Week 18 scores, 1 sided test for Treatment Group Superiority; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Parent Child Interaction Therapy vs Wait List Control; Comparison of DPICS Positive Skills between Week 18 scores, 1 sided test for Treatment Group Superiority. Data transformed using a square root transformation; Test type: Superiority; p < .001, t-test, 1 sided — No adjustment for multiple comparisons

8. Secondary Outcome: Parental Stress Index Score
Description: Parental Stress Index-4 Short Form (PSI):Total Stress Scale, total of subscales, range 36-180, higher indicating more parental stress. Defensive Responding, range 7-35. Lower scores indicate higher defensive responding from parents. Parental Distress, range 12-60. Higher scores indicate more parental stress. Parent-Child Dysfunctional Interaction subscale, range 12-60. Higher scores indicate parents feel their child is not meeting their expectations when interacting. Difficult Child, range is 12-60. Higher scores indicate that parents view their child to be difficult to parent.
Time Frame: Week 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Child Interaction Therapy | Wait List Control
Number analyzed (Participants) | 10 | 9
units on a scale
  PSI DR | 18.80 (7.15) | 19.56 (5.41)
  Parent Distress Subscale Score | 31.30 (11.20) | 31.44 (8.93)
  Parent-Child Dysfunctional Interaction Subscale Sc | 31.30 (9.26) | 28.78 (11.65)
  Difficult Child Subscale Score | 41.30 (10.67) | 41.11 (8.45)
  Total Stress | 103.90 (28.18) | 101.33 (24.77)

ADVERSE EVENTS:
Time Frame: The time frame that information on adverse events was collected depended on which treatment assignment was made. For individuals who were assigned to immediate PCIT training, adverse event data was collected over a period of 18 - 30 weeks, dependent on the subject's ability to schedule training. For individuals on the wait list for PCIT, adverse event data was collected over a period of 30 - 48 weeks, dependent on the subject's ability to schedule training.
Arm/Group | Parent Child Interaction Therapy | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No